CLINICAL TRIAL: NCT04030013
Title: "Outcome of Diabetes Education Among Renal Transplant Recipients With New Onset Diabetes After Transplantation (NODAT)"
Acronym: NODAT-ES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Nashwa Othman, Senior specialist diabetes educator, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RA 2014-049
Record Dates: First submitted 2017-03-15; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: New Onset Diabetes After Transplant; Diabetes Mellitus
Keywords: renal; diabetes; outcome; transplant; Education
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group education for 2 years (Active Comparator): Patients who will receive structured diabetes education in groups , Group 1
  Interventions: Other: group education
- One to one education for 2 years (Active Comparator): Patients who will receive one to one structured diabetes education, Group 2
  Interventions: Other: group education
- Control group without structured education (No Intervention): Patients who will not receive structured diabetes education, Group 3

INTERVENTIONS:
Other: group education — All patients of group 1 and 2 will receive intensive education for 3-4 months, then refreshment session every 3 months for 2 years. Initially, patient data will be collected through 3 types of forms: patient identification form, metabolic control parameters form and diabetes self-care scale questionnaire; then every 6 months metabolic parameters and diabetes self-care scale questionnaire will be reassessed.
  Other Names: one to one; conventional education
  Arms: Group education for 2 years; One to one education for 2 years

SUMMARY:
Introduction:

Diabetes is a chronic disease that requires lifelong self care behavior. Successful treatment of chronic diseases is closely associated with the education of both patients and their relatives. Patient education is one of the most important responsibilities of diabetes nurse educators. In the management of diabetes, helping patients to improve their health and quality of life is considered an important aspect of diabetes self-care education. Solid organ transplantation is now the standard of care for end-stage organ failure. New-onset diabetes mellitus after solid organ transplantation (NODAT) has emerged as an increasingly important determinant of outcomes and survival in transplant recipients. Patient education and self-management are crucial for ensuring successful outcome post transplantation. No adequate studies concerning education of diabetic renal transplants.

Aim of the work: The aim of this work is to evaluate the effect of diabetes education given to renal transplant recipients with new onset diabetes after transplantation (NODAT) on their self-care activities and metabolic control variables and reversibility of the present chronic diabetic complications.

Patients and methods:

The study will involve 210 diabetic renal transplant patients (NODAT) who will be referred from Hamed Al-Essa organ transplant center to Dasman Diabetes Institute. These patients will be sub-divided into three subgroups: patients who will receive group education (n=70) will represent group1, patients who will receive one to one education (n=70) will represent group 2, while those who will receive the conventional (not structured) education program will serve as control group 3(n= 70). All patients of group 1 and 2 will receive intensive education for 3-4 months, then refreshment session every 3 months for 2 years. Initially, patient data will be collected through 3 types of forms: patient identification form, metabolic control parameters form and diabetes self-care scale questionnaire; then every 6 months metabolic parameters and diabetes self-care scale questionnaire will be reassessed.

Expected outcome: Patient education given to transplant recipients with NODAT could affect patients' self-care activities, metabolic control positively and possibly help in reversal of chronic diabetic complications

DETAILED DESCRIPTION:
The research population will include organ transplant recipients with NODAT who are followed up in Hamed AL-Essa organ transplant centre of Kuwait and who will meet the eligibility criteria. Two hundred and ten diabetic renal transplant recipients will be enrolled in this prospective randomised controlled study. Patients who fulfil the following criteria will be included in the study: 1) transplant duration more than 6 months; 2) being an outpatient; 3) not having any psychiatric history of illness; 4) written consent to participate in the research; and 5) age of diabetic patients more than 21 years . We will exclude paediatrics (bellow 21 years) and mentally abnormal patients. Ethical principles of the research Written permission will be received from the institutions where the research will be carried out. Information form including the aim and scope of the research will be submitted to Ethical Committees of both ministry of health (MOH) of Kuwait and Dasman Diabetes Institute.

Data collection tools

Patient identification form:

This form will include information about the patient's identifying characteristics such as age, gender, education status and disease-related information such as duration of the disease and the treatments management of diabetes.

Metabolic control parameters form:

This form will include patient's metabolic control variables such as HbA1c, lipids (Total cholesterol, triglyceride, high-density lipoprotein (HDL), low-density lipoprotein (LDL), renal and liver function tests. Metabolic control parameters will be measured in Hamed Al-Essa organ transplantation center (OTC) outpatient clinic and will be sent with each patient to Dasman Diabetes Institute within one week of patient evaluation for starting educational program.

Blood pressure, height, weight, body mass index and waist circumference of patients will be measured and recorded by the researcher each time by using the same measurement device and method. Patients' waist circumferences will be measured midway between costal margin and iliac crests by a measuring tape in standing position, over underwear and after slight expiration.

Diabetes self-care scale (DSCS) The Arabic translated 24-items scale- developed in English by Lee and Fisher(41) which measures the self care of patients with diabetes -will be applied to patients before and after the education program.

Data collection method In the pretest phase of the research, patients will be given a patient identification form, metabolic control parameters form and a DSCS. The forms will be completed within15-25 minutes by the patients in the presence of the researcher. Telephone numbers and addresses of patients will be taken for proper communication if needed.

Patient education Group education sessions will be carried out in special halls in Dasman Diabetes Institute (DDI) after proper coordination with the randomly selected patients (group 1) (6-10 patients in each education group). Patients of one to one education group (group 2) will receive education sessions individually in closed education clinics of DDI. The first session will last for 60 minutes then the next sessions will last for 30 minutes. The content of education will be repeated entirely or partly by the researcher according to each patient's needs. Mixed education techniques such as description, question and answer techniques will be used as an education method and feedback will be stimulated trying to enable patients to understand their self-care management independently. Refreshment education sessions will be delivered every 3 months later on till the end of the study.

Regarding patients of the third group (control group), each patient will receive the conventional (non-structured) education program in their mother hospital (OTC).

ELIGIBILITY:
Inclusion Criteria:

* 1) transplant duration more than 6 months; 2) being an outpatient; 3) not having any psychiatric history of illness; 4) written consent to participate in the research; and 5) age of diabetic patients more than 21 years

Exclusion Criteria:

* pediatrics (bellow 21years) and mentally abnormal patients.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-07

PRIMARY OUTCOMES:
Evaluate the effect of diabetes education given to renal transplant recipients with new onset diabetes after transplantation . | For 2 years from the time of enrolment
  Positive metabolic control and self-care diabetes management

SECONDARY OUTCOMES:
comparison of type of diabetes education | For 2 years from the enrolment
  Comparison between one to one vs. group education

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa F Othman, MD PhD, Principal Investigator — Senior diabetes educator in Dasman Diabetes Institute; Osama A Gheith, MD PhD, Study Director — Consultant nephrologist, Hamed Al-Essa organ transplnat center
Locations (1):
- Dasman diabetes institute, Kuwait City, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No